CLINICAL TRIAL: NCT00191906
Title: A Randomized, Double-Blind, Crossover Comparison of Atomoxetine and Placebo in Child Outpatients With Attention-Deficit/Hyperactivity Disorder, Reading Disorder, or Comorbid Attention-Deficit/Hyperactivity Disorder and Reading Disorder.
Brief Title: Comparison of Atomoxetine and Placebo in Children With Attention-Deficit/Hyperactivity Disorder (ADHD) and/or Reading Disorder (RD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7955; B4Z-MC-LYCK (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2010-04-06 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Attention Deficit Hyperactivity Disorder; Reading Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dyslexia | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Atomoxetine first, then Placebo (Experimental): Atomoxetine, 1.2 mg/kg/day, by mouth (PO) for 4 weeks, 2 week washout period and cross-over to placebo, every day (QD), PO for 4 weeks
  Interventions: Drug: Atomoxetine Hydrochloride; Drug: placebo
- Placebo first, then Atomoxetine (Experimental): Placebo, every day (QD), by mouth (PO) for 4 weeks, 2 week washout period and cross-over to atomoxetine 1.2 mg/kg/day, PO for 4 weeks
  Interventions: Drug: Atomoxetine Hydrochloride; Drug: placebo
- Normal Control (No Intervention): Normal controls were children selected from the general population. The normal control was matched (have same proportion) by sex (male/female) and by age (have same age range) as the study population.
- Reading Disordered Control (No Intervention): The reading disordered control group is comprised of children with reading disorder who receive standard remedial teaching therapy.

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride — Atomoxetine, 1.2 mg/kg/day, by mouth (PO)
  Other Names: LY139603; Strattera
  Arms: Atomoxetine first, then Placebo; Placebo first, then Atomoxetine
Drug: placebo — Placebo, every day (QD), by mouth (PO)
  Arms: Atomoxetine first, then Placebo; Placebo first, then Atomoxetine

SUMMARY:
To test the hypothesis that a 4 week treatment with atomoxetine is more effective than placebo in patients with combined type Attention Deficit/Hyperactivity Disorder (ADHD), patients with only Reading Disorder, and patients with combined type ADHD and Reading Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis with Attention Deficit Hyperactivity Disorder and/or Reading Disorder

Exclusion Criteria:

* Patients with Conduct Disorder
* Patients who have a history of Bipolar I or II Disorder, psychosis, or Pervasive Development Disorder.
* Patients who have a current diagnosis of Vocal Tic Disorder, Obsessive Compulsive Disorder, Major Depressive Disorder, Post Traumatic Stress Disorder, Anxiety Disorder, and certain other learning disorders.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 . Mon-Fri 9AM - 5PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent, Belgium
- Netherlands (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Almere Stad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Breda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vught

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- [Derived] de Jong CG, Van De Voorde S, Roeyers H, Raymaekers R, Allen AJ, Knijff S, Verhelst H, Temmink AH, Smit LM, Rodriques-Pereira R, Vandenberghe D, van Welsen I, ter Schuren L, Al-Hakim M, Amin A, Vlasveld L, Oosterlaan J, Sergeant JA. Differential effects of atomoxetine on executive functioning and lexical decision in attention-deficit/hyperactivity disorder and reading disorder. J Child Adolesc Psychopharmacol. 2009 Dec;19(6):699-707. doi: 10.1089/cap.2009.0029. PMID 20035588
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Period I: screening/washout (89 patients screened, 13 screen-failures;45 controls screened). Period II (Visits 2-5): patients received treatment for 4 weeks and then underwent 2-week washout period after which they crossed over to receive the alternate treatment for 4 additional weeks. Period III (Visits 6-12): optional open-label (1 country only).
Groups:
- Atomoxetine First, Then Placebo: Atomoxetine 1.2 mg/kg/day, by mouth for 4 weeks, 2 week washout period and then cross-over to placebo, every day, by mouth for 4 weeks.
- Placebo First, Then Atomoxetine: Placebo every day, by mouth for 4 weeks, 2 week washout period and then cross-over to atomoxetine 1.2 mg/kg/day, by mouth for 4 weeks.
- Normal Control: Untreated normal controls were children selected from the general population. The normal control was matched (have same proportion) by sex (male/female) and by age (have same age range) as the study population.
- Reading Disordered Control: Untreated reading disordered control group was comprised of children with reading disorder who received standard remedial teaching therapy.
Period: Study Period II
Arm/Group | Atomoxetine First, Then Placebo | Placebo First, Then Atomoxetine | Normal Control | Reading Disordered Control
Started | 39 | 37 | 27 | 18
Completed | 39 | 32 | 26 | 18
Not Completed | 0 | 5 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0
Not completed — Parent/Caregiver Decision | 0 | 1 | 0 | 0
Not completed — Entry Criteria Exclusion | 0 | 0 | 1 | 0
Period: Study Period III
Arm/Group | Atomoxetine First, Then Placebo | Placebo First, Then Atomoxetine | Normal Control | Reading Disordered Control
Started | 14 (These are patients who continued in optional open-label period (1 country). All received atomoxetine) | 11 (These are patients who continued in optional open-label period (1 country). All received atomoxetine) | 0 | 0
Completed | 9 | 7 | 0 | 0
Not Completed | 5 | 4 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Parent/Caregiver Decision | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine First, Then Placebo: Atomoxetine 1.2 mg/kg/day for 4 weeks, 2 week washout, and then placebo for 4 weeks
- Placebo First, Then Atomoxetine: Placebo for 4 weeks, 2 week washout, and then atomoxetine 1.2 mg/kg/day for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Atomoxetine First, Then Placebo | Placebo First, Then Atomoxetine | Normal Control | Reading Disordered Control | Total
Number analyzed (Participants) | 39 | 37 | 27 | 18 | 121
Age Continuous [Mean (Standard Deviation); unit: years] | 10.0 (1.34) | 9.9 (1.25) | 9.9 (1.01) | 10.6 (0.99) | 10.0 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 10 | 5 | 38
  Male | 26 | 27 | 17 | 13 | 83
Region of Enrollment [Number; unit: participants]
  Belgium | 18 | 15 | 0 | 16 | 49
  Netherlands | 21 | 22 | 27 | 2 | 72
Study Arm - Diagnosis [Number; unit: participants]
  ADHD-Combined Type | 13 | 15 | 0 | 0 | 28
  Reading Disorder | 11 | 12 | 0 | 18 | 41
  ADHD-Combined Type + Reading Disorder | 15 | 10 | 0 | 0 | 25
  No Disorder | 0 | 0 | 27 | 0 | 27

OUTCOME MEASURES:

1. Primary Outcome: Stop Signal Reaction Time (SSRT) as Derived From the Stop Signal Reaction Time Paradigm
Description: SSRT measures response execution (go trials) and response inhibition (stop trials). Go trials consist of stimulus (airplane). Child to press response button corresponding to direction airplane is pointing. Stop trials consist of go trial and audible stop signal. Initial delay between go trial and stop signal = 250 msec. If child succeeded in inhibiting response, delay on next stop trial increased by 50 msec, otherwise, delay decreased by 50 msec. SSRT = subtract mean delay from mean go signal reaction time. Lower scores mean better ability to suppress response when presented with stop signal.
Time Frame: Baseline and Week 4 of initial therapy and Week 4 of crossover therapy
Population: All efficacy information is summarized and/or presented in data listings based on the Safety sample: Includes all patients who were randomized to double-blind treatment and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Groups:
- Atomoxetine: Atomoxetine, 1.2 mg/kg/day, by mouth for 4 weeks.
- Placebo: Placebo, daily, by mouth for 4 weeks.
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 71 | 76
milliseconds (msec)
  ADHD-Combined Type | 299.90 (13.29) | 308.82 (14.53)
  Reading Disorder | 265.61 (14.24) | 260.51 (16.02)
  ADHD-C + Reading Disorder | 277.38 (13.80) | 292.53 (15.46)
  Overall | 280.97 (7.96) | 287.29 (8.84)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Least Squares Mean (LSMean) values were calculated from the measurements taken at baseline and at the end of each 4 week therapy period; Test type: Superiority or Other; p = 0.504, Repeated Measures — P-value for Overall. No adjustments for multiple comparisons - not applicable. All statistical tests were performed using a 0.05 significance level; Repeated measures model including terms for baseline, study arm, treatment sequence, visit, treatment, and treatment-by-study-arm interaction

2. Secondary Outcome: Change From Baseline in Mean Stop Signal Reaction Time Comparison of ADHD-C to Normal Control Group in >=10 Year Old Subset
Description: as for outcome 1
Time Frame: Baseline and 4 weeks of therapy
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- ADHD-C: atomoxetine-treated Attention-Deficit/Hyperactivity Disorder-Combined Type
Arm/Group | ADHD-C | Normal Control
Number analyzed (Participants) | 5 | 8
milliseconds | 7.95 (48.21) | 11.22 (62.77)
Statistical Analysis 1: Comparison: ADHD-C vs Normal Control; ANCOVA model with baseline value, study arm as covariates for ADHD-C versus Normal controls; Test type: Superiority or Other; p = 0.970, ANCOVA — There were no adjustments for multiple comparisons - not applicable. All statistical tests were performed using a 0.05 significance level

3. Secondary Outcome: Change From Baseline in Mean Stop Signal Reaction Time Comparison of ADHD-C+RD and RD to Reading Disordered Control Group in >=10 Year Old Subset
Description: as for outcome 1
Time Frame: Baseline and 4 weeks of therapy
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- ADHD-C+RD: atomoxetine-treated Comorbid Attention-Deficit/Hyperactivity Disorder-Combined Type + Reading Disorder
- Reading Disorder: atomoxetine-treated Reading Disorder
Arm/Group | ADHD-C+RD | Reading Disorder | Reading Disordered Control
Number analyzed (Participants) | 16 | 13 | 14
milliseconds | -0.25 (53.41) | -34.0 (33.91) | 0.05 (24.08)
Statistical Analysis 1: Comparison: ADHD-C+RD vs Reading Disordered Control; ANCOVA model with baseline value, study arm as covariates for ADHD-C+RD versus RD controls; Test type: Superiority or Other; p = 0.579, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Reading Disorder vs Reading Disordered Control; ANCOVA model with baseline value, study arm as covariates for RD versus RD controls; Test type: Superiority or Other; p = 0.144, ANCOVA — There were no adjustments for multiple comparisons - not applicable. All statistical tests are performed using a 0.05 significance level

4. Secondary Outcome: Lexical Decision Task Mean Reaction Time: Correct Words
Description: Measure of reaction time to identify whether a word displayed on a computer is a real or correct word versus a pseudo word. During the performance of the lexical decision task that was presented on a computer, the reaction times and accuracy of responses were measured. Data presented are the mean reaction times over the 4 weeks of each therapy for identifying correct words correctly.
Time Frame: Baseline and Week 4 of initial therapy and Week 4 of crossover therapy
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 68 | 73
milliseconds
  ADHD-Combined Type | 1182.9 (50.23) | 1291.9 (38.13)
  Reading Disorder | 1172.4 (51.75) | 1198.6 (40.24)
  ADHD-C + Reading Disorder | 1201.9 (51.22) | 1305.9 (39.43)
  Overall | 1185.7 (29.49) | 1265.5 (22.61)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.005, Repeated Measures — P-value for Overall. There were no adjustments for multiple comparisons - not applicable. All statistical tests were performed using a 0.05 significance level; Repeated measures model including terms for baseline, study arm, treatment sequence, visit, treatment, and treatment by study-arm-interaction

5. Secondary Outcome: Lexical Decision Task Mean Reaction Time: Pseudo Words
Description: Measure of reaction time to identify whether a word displayed on a computer is a pseudo word versus a real or correct word. During the performance of the lexical decision task that was presented on a computer, the reaction times and accuracy of responses were measured. Data presented are the mean reaction times over the 4 weeks of each therapy for identifying pseudo words correctly.
Time Frame: Baseline and Week 4 of initial therapy and Week 4 of crossover therapy
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 68 | 73
milliseconds
  ADHD-Combined Type | 1403.0 (63.72) | 1475.4 (50.08)
  Reading Disorder | 1365.0 (65.62) | 1412.2 (52.90)
  ADHD-C + Reading Disorder | 1426.1 (64.83) | 1487.0 (51.73)
  Overall | 1398.0 (37.33) | 1458.2 (29.63)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.097, Repeated Measures — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Working Memory by Corsi Block Tapping Test (CBTT)
Description: Measures the visuo-spatial working memory span, and corresponds to the longest sequence of blocks that has been reproduced correctly at least once. Scores can range from 3 to 8, with the higher score indicating better function.
Time Frame: Baseline and Week 4 of initial therapy and Week 4 of crossover therapy
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: blocks correctly sequenced
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 69 | 73
blocks correctly sequenced
  ADHD-Combined Type | 5.29 (0.22) | 4.98 (0.21)
  Reading Disorder | 5.50 (0.23) | 5.14 (0.23)
  ADHD-C + Reading Disorder | 5.92 (0.23) | 5.29 (0.23)
  Overall | 5.57 (0.13) | 5.14 (0.13)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.003, Repeated Measures — [p-value comment as in outcome 4, analysis 1]; Repeated measures model including terms for study arm, treatment sequence, treatment, and treatment-by-study-arm interaction

7. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version: Investigator-Administered and Scored - Total Score
Description: Measures the 18 symptoms contained in the DSM-IV diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total score is the sum of the scores on the 18 items and range from 0 to 54.
Time Frame: Baseline and Week 4 of initial therapy and Week 4 of crossover therapy
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 46 | 47
units on a scale
  ADHD-Combined Type | 30.86 (2.14) | 35.20 (1.78)
  ADHD-Combined Type + Reading Disorder | 22.44 (2.38) | 35.17 (2.07)
  Overall | 26.65 (1.60) | 35.18 (1.34)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated Measures — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version: Investigator-Administered and Scored - Inattention Subscale
Description: Measures the degree of inattention symptoms based on answers to 9 items. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often), for a total Inattention Subscale score range of 0 to 27.
Time Frame: Baseline and Week 4 of initial therapy and Week 4 of crossover therapy
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 46 | 47
units on a scale
  ADHD-Combined Type | 15.27 (1.09) | 17.82 (0.93)
  ADHD-Combined Type + Reading Disorder | 12.25 (1.22) | 18.28 (1.09)
  Overall | 13.76 (0.82) | 18.05 (0.70)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated Measures — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version: Investigator-Administered and Scored - Hyperactivity-Impulsivity Subscale
Description: Measures the degree of hyperactivity-impulsivity symptoms, based on answers to 9 items. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often) for a total Hyperactivity-Impulsivity Subscale score of 0 to 27.
Time Frame: Baseline and Week 4 of initial therapy and Week 4 of crossover therapy
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 46 | 47
units on a scale
  ADHD-Combined Type | 15.51 (1.14) | 17.24 (0.96)
  ADHD-Combined Type + Reading Disorder | 10.32 (1.27) | 17.03 (1.12)
  Overall | 12.91 (0.85) | 17.13 (0.73)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated Measures — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version: Investigator-Administered and Scored - Total T-Score
Description: Measures the 18 symptoms contained in the DSM-IV diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total score is computed as the sum of the scores on each of the 18 items. Total score is the sum of the scores on the 18 items and range from 0 to 54. Total T-score = (Total Score - 50)/10. Total T-score ranges from -5 (low severity) to 0.4 (high severity).
Time Frame: Baseline and Week 4 of initial therapy and Week 4 of crossover therapy
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-Score of units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 46 | 47
T-Score of units on a scale
  ADHD-Combined Type | -1.91 (0.21) | -1.48 (0.18)
  ADHD-Combined Type + Reading Disorder | -2.76 (0.24) | -1.48 (0.21)
  Overall | -2.34 (0.16) | -1.48 (0.13)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated Measures — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 1, analysis 1]

11. Secondary Outcome: Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Improvement Scale
Description: Measures total improvement (or worsening) of a patient's ADHD symptoms from the beginning of treatment (1=very much improved, 7=very much worsened).
Time Frame: 4 week therapy endpoint
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 47 | 52
units on a scale
  ADHD-Combined Type | 3.69 (0.24) | 3.70 (0.23)
  ADHD-Combined Type + Reading Disorder | 2.98 (0.24) | 3.76 (0.24)
  Overall | 3.34 (0.17) | 3.73 (0.16)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.094, Repeated Measures — [p-value comment as in outcome 4, analysis 1]; Repeated measures model including terms for study arm, treatment sequence, visit, treatment, and treatment-by-study-arm interaction

12. Secondary Outcome: Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Severity Scale
Description: Measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: 4 week therapy endpoint
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 47 | 52
units on a scale
  ADHD-Combined Type | 4.05 (0.21) | 3.73 (0.19)
  ADHD-Combined Type + Reading Disorder | 3.65 (0.21) | 4.34 (0.20)
  Overall | 3.85 (0.14) | 4.04 (0.13)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.312, Repeated Measures — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 1, analysis 1]

13. Secondary Outcome: Change From Baseline in Phonological Task Mean Reaction Time Comparison of ADHD-C to Normal Control Group in >=10 Year Old Subset: Pseudohomophones
Description: Measure of reaction time in determining whether the stimulus sounds like a real word ('yes' response) or not ('no' response) using pseudohomophones and pseudo words. Data presented here are for reaction time to identifying psuedohomophones correctly.
Time Frame: Baseline and 4 weeks of therapy
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | ADHD-C | Normal Control
Number analyzed (Participants) | 5 | 6
milliseconds | -230.40 (239.43) | -339.17 (176.32)
Statistical Analysis 1: Comparison: ADHD-C vs Normal Control; ANCOVA model with baseline value, study arm as covariates for ADHD-C versus normal controls; Test type: Superiority or Other; p = 0.508, ANCOVA — [p-value comment as in outcome 2, analysis 1]

14. Secondary Outcome: Change From Baseline in Phonological Task Mean Reaction Time Comparison of ADHD-C to Normal Control Group in >=10 Year Old Subset: Pseudo Words
Description: Measure of reaction time in determining whether the stimulus sounds like a real word ('yes' response) or not ('no' response) using pseudo homophones and pseudo words. Data presented here are for reaction time to identifying pseudo words correctly.
Time Frame: Baseline and 4 weeks of therapy
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | ADHD-C | Normal Control
Number analyzed (Participants) | 5 | 6
milliseconds | -523.20 (524.36) | -536.00 (303.27)
Statistical Analysis 1: Comparison: ADHD-C vs Normal Control; ANCOVA model with baseline value, study arm as covariate for ADHD-C versus normal controls; Test type: Superiority or Other; p = 0.769, ANCOVA — [p-value comment as in outcome 2, analysis 1]

15. Secondary Outcome: Change From Baseline in Phonological Task Mean Reaction Time Comparison of ADHD-C+RD and RD to Reading Disordered Control Group in >=10 Year Old Subset: Pseudohomophones
Description: Measure of reaction time in determining whether the stimulus sounds like a real word ('yes' response) or not ('no' response) using pseudo homophones and pseudo words. Data presented here are for reaction time to identifying psuedohomophones correctly.
Time Frame: Baseline and 4 weeks of therapy
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- ADHD-C+ RD: atomoxetine-treated Comorbid Attention-Deficit/Hyperactivity Disorder-Combined Type + Reading Disorder
Arm/Group | ADHD-C+ RD | Reading Disorder | Reading Disordered Control
Number analyzed (Participants) | 16 | 13 | 14
milliseconds | -170.81 (243.33) | -241.00 (317.47) | -254.86 (266.46)
Statistical Analysis 1: Comparison: ADHD-C+ RD vs Reading Disordered Control; ANCOVA model with baseline value, study arm as covariates for ADHD-C+RD versus RD controls; Test type: Superiority or Other; p = 0.302, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Reading Disorder vs Reading Disordered Control; ANCOVA model with baseline value, study arm as covariate for RD versus RD controls; Test type: Superiority or Other; p = 0.663, ANCOVA — [p-value comment as in outcome 2, analysis 1]

16. Secondary Outcome: Change From Baseline in Phonological Task Mean Reaction Time Comparison of ADHD-C+RD and RD to Reading Disordered Control Group in >=10 Year Old Subset: Pseudo Words
Description: Measure of reaction time in determining whether the stimulus sounds like a real word ('yes' response) or not ('no' response) using pseudo homophones and pseudo words. Data presented here are for reaction time to indentifying pseudo words correctly.
Time Frame: Baseline and 4 weeks of therapy
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- ADHD-C+RD: atomoxetine-treated Attention-Deficit/Hyperactivity Disorder-Combined Type + Reading Disorder
Arm/Group | ADHD-C+RD | Reading Disorder | Reading Disordered Control
Number analyzed (Participants) | 16 | 13 | 14
milliseconds | -113.06 (432.68) | -213.00 (512.33) | -368.14 (422.42)
Statistical Analysis 1: Comparison: ADHD-C+RD vs Reading Disordered Control; ANCOVA model with baseline value, study arm as covariate for ADHD-C+RD versus RD controls; Test type: Superiority or Other; p = 0.070, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Reading Disorder vs Reading Disordered Control; ANCOVA model with baseline value, study arm as covariate for RD versus RD controls; Test type: Superiority or Other; p = 0.179, ANCOVA — [p-value comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Groups:
- As Randomized Placebo (Crossover): Patients in either Crossover Period receiving Placebo
- As Randomized Atomoxetine (Crossover): Patients in either Crossover Period receiving Atomoxetine
- Open Label Atomoxetine: Patients in the Open Label extension receiving Atomoxetine
Arm/Group | As Randomized Placebo (Crossover) | As Randomized Atomoxetine (Crossover) | Open Label Atomoxetine
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/74 | 0/25
Other Adverse Events (participants affected / at risk) | 28/76 | 35/74 | 24/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | As Randomized Placebo (Crossover) (N=76) | As Randomized Atomoxetine (Crossover) (N=74) | Open Label Atomoxetine (N=25)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Mydriasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual disturbance (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 6 (7) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (7) | 3 (4)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (5) | 2 (3)
Fatigue (General disorders) | 2 (2) | 9 (11) | 4 (4)
Feeling abnormal (General disorders) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0)
Peripheral coldness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 6 (6) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 10 (11) | 10 (10) | 8 (9)
Poor quality sleep (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Apathy (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Eating disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Fear (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Negativism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Job dissatisfaction (Social circumstances) | 1 (1) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 2 (2) | 2 (3) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days